CLINICAL TRIAL: NCT05691296
Title: The Monitoring and Intervention of Refractive Changes in Children and Teenagers in Tianjin
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Tianjin myopia Intervention
Record Dates: First submitted 2022-12-25; First posted 2023-01-20 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Myopia; High Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home-school training group (Experimental): There was a Letter Chart Accomodative Rock Training for accommodation facility at home and school everyday. This training usually lasted 2 minutes each time.
  Interventions: Behavioral: Home training; Behavioral: School training
- School training group (Experimental): There was a Letter Chart Accomodative Rock Training for accommodation facility only at school everyday. This training usually lasted 2 minutes each time.
  Interventions: Behavioral: School training
- No training group (No Intervention): There was no such treatment for students.

INTERVENTIONS:
Behavioral: Home training — Letter Chart Accomodative Rock Training for 2 minutes each time
  Arms: Home-school training group
Behavioral: School training — Letter Chart Accomodative Rock Training for 2 minutes each time
  Arms: Home-school training group; School training group

SUMMARY:
The study aimed to collect multi-factor information on school-age children with pre-clinical myopia, and to identify the initial factors and warning signs of myopia.

DETAILED DESCRIPTION:
The incidence of myopia is high in China. At present, the mechanism of myopia is unclear, and the main theories are genetic and environmental aspects. Many factors may affect the occurrence and development of myopia in students, such as ocular biological parameters, peripheral refractive state, differences in binocular vision function, eye habits, and outdoor time. In this study, the multi-factor information on pre-clinical myopia in school-age children was collected to find out the initial factors and warning signals of myopia.

ELIGIBILITY:
Inclusion Criteria:

* All students in grades 1 to 4
* Can cooperate with the examination of students

Exclusion Criteria:

* Obvious strabismus and amblyopia
* Eye diseases that affect vision, such as congenital cataracts, glaucoma, and retinal diseases
* History of ocular surgery

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4000 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of new-onset myopia | Through study completion, an average of 1 year
  The number of new children with myopia was counted
The changes of refractive error | Every 6 months, up to 3 years
  The changes of refractive error between visit time and baseline which was obtained with a computer refractometer.
The changes of axial length | Every 6 months, up to 3 years
  The axial length was measured by a biological measuring instrument.

CONTACTS AND LOCATIONS:
Locations (1):
- Tiajin Eye Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Background] Jonas JB, Ang M, Cho P, Guggenheim JA, He MG, Jong M, Logan NS, Liu M, Morgan I, Ohno-Matsui K, Parssinen O, Resnikoff S, Sankaridurg P, Saw SM, Smith EL 3rd, Tan DTH, Walline JJ, Wildsoet CF, Wu PC, Zhu X, Wolffsohn JS. IMI Prevention of Myopia and Its Progression. Invest Ophthalmol Vis Sci. 2021 Apr 28;62(5):6. doi: 10.1167/iovs.62.5.6. PMID 33909032